CLINICAL TRIAL: NCT04836715
Title: Prevalence of Visual Dysfunction in Persons With Parkinson's Disease and Other Neurological Disorders
Brief Title: Prevalence of Visual Dysfunction in Neurological Disorders
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202100649
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease; Other Neurological Disorders; Healthy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Parkinson's Disease: Individuals with idiopathic Parkinson's Disease and no other neurological disease
- Other Neurological Disorders: Individuals with one neurological disorder other than Parkinson's Disease (e.g. Multiple Sclerosis, Amyotrophic Lateral Sclerosis, Traumatic Brain Injury, Parkinsonism)
- Healthy: Individuals without any neurological disorder

SUMMARY:
The objective is to determine the prevalence of visual dysfunction in People with Parkinson's Disease (PwP). The investigators will administer the: Visual Impairment in Parkinson's Disease Screen and Revised-Self-Report Assessment of Functional Visual Performance. Patients seen at Fixel Institute and their caregivers will be invited to participate. Responses to the 2 questionnaires will help determine prevalence rates of visual dysfunction in PwP compared to those both with and without other neurological conditions.

DETAILED DESCRIPTION:
The purpose of this study is to identify the prevalence of visual dysfunction among Persons with Parkinson's Disease, compared to other neurological conditions and controls without neurological conditions.

Data will be collected anonymously via RedCap. Patients seen at the Fixel Institute that have consented to be contacted regarding research opportunities will be recruited via blast email and advertisement in our Institute's monthly newsletter, the Movement Messenger. The email and newsletter will contain a link for participation in surveys within RedCap so the surveys can be completed anonymously at home. Participation will be completely voluntary and responses will be recorded anonymously. Data will include responses to the following: screening questions, the VIPDQ (Visual Impairment in PD Questionnaire), and the R-SRAFVP (Revised-Self-Report Assessment of Functional Visual Performance).

The investigators will calculate the prevalence of visual impairment (from the VIPDQ) and dysfunction in performance of daily activities (from the R-SRAFVP) for PwP and compare this to the prevalence occurring in other neurological populations as well as the population without any neurological conditions. Other data are collected so the investigators can then evaluate potential confounds or covariates. To ensure statistical methods are accurate, a statistician will be consulted.

ELIGIBILITY:
Inclusion Criteria:

* Persons with Parkinson's Disease: Confirmed diagnosis of Parkinson's Disease without presence of any other neurological condition.
* Persons without Parkinson's Disease (Controls): No previous diagnosis of any neurological condition
* Persons with a single other neurological disorder (Neuro Controls): Confirmed diagnosis of other neurological condition (e.g. ALS, multiple sclerosis, essential tremor, ataxia, etc).

Exclusion Criteria:

* Children (ages younger than 18 years of age)
* Persons with more than one diagnosed neurological condition.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Persons with Parkinson's Disease
  2. Persons without a Neurological Condition (Controls)
  3. Persons with Other Neurological Conditions (e.g. ALS, TBI, MS, CBT/CBS, MSA, PSP, MCI, etc).
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Visual Dysfunction | 1 day
  Determined from VIPDQ: (with the highest and lowest scores on the VIPD-Q Score). Answers are given on a 4-point Likert scale ranging from "never have problems" to "daily problems"
Functional Visual Performance | 1 day
  Determined from R-SRA FVP: SRAFVP %

OTHER OUTCOMES:
Correlations between Visual Dysfunction and Functional Visual Performance | 1 day
  Correlation Coefficient: VIPDQ score and SRAFVP % will be analyzed statistically to report correlation coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Nicole J Tester, PhD, MOT, OTR/L, MSCS, Principal Investigator — University of Florida/UF Health Rehab
Locations (2):
- United States (2):
  - UF Health Rehab - Fixel Institute, Gainesville, Florida
  - University of Florida, Gainesville, Florida